CLINICAL TRIAL: NCT05854602
Title: The Relative Effects of Three Parent-Intervention Components to Reduce Children's Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Karen Rienks, PhD Candidate, University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: VI.Vidi.201.065 - Study 5
Record Dates: First submitted 2023-04-19; First posted 2023-05-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Anxiety
Keywords: Anxiety; Children; Parents; Prevention; Intervention
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: A Factorial Experiment with 34 conditions
Who Masked: Participant
Masking Description: Participants and researchers will be blinded to condition at enrolment and baseline assessment.
  Randomization takes place after baseline assessment (T0), by drawing a number (1-34, corresponding to condition 1-34) from a sealed envelope, by a researcher who has no contact with any of the study participants.
  Care providers cannot be blinded to participants' condition. At T2/4/6/12, Participants will be blinded to the conditions that exist in the study, but are aware of whether they received one or more intervention components.
  Independent researchers and clinicians blinded to participants' condition and timepoint (T0/6/12) will code video recordings of the parent-child interaction task and parental stories about children's anxiety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (34):
- Condition 1: 000 (No Intervention): Families in this condition will not receive any of the intervention components during study period (T0-T2, T2-T4, T4-T6). Target n = 35.
- Condition 2: 0A0 (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A
- Condition 3: 00A (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A
- Condition 4: 0AB (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 5: 0AC (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 6: 0B0 (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B
- Condition 7: 00B (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B
- Condition 8: 0BA (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 9: 0BC (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 10: 0C0 (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component C
- Condition 11: 00C (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component C
- Condition 12: 0CA (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 13: 0CB (Experimental): This intervention condition received no intervention from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 14: A00 (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A
- Condition 15: A0B (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 16: A0C (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 17: AB0 (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 18: ABC (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C
- Condition 19: AC0 (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 20: ACB (Experimental): This intervention condition received Component A from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C
- Condition 21: B00 (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B
- Condition 22: B0A (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 23: B0C (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 24: BA0 (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B
- Condition 25: BAC (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and Component C from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C
- Condition 26: BC0 (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 27: BCA (Experimental): This intervention condition received Component B from baseline (T0) to the second measurement point two weeks later (T2), Component C from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C
- Condition 28: C00 (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component C
- Condition 29: C0A (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 30: C0B (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), no intervention from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 31: CA0 (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component C
- Condition 32: CAB (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), Component A from T2 to two weeks later (T4), and Component B from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C
- Condition 33: CB0 (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and no intervention from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component B; Behavioral: Component C
- Condition 34: CBA (Experimental): This intervention condition received Component C from baseline (T0) to the second measurement point two weeks later (T2), Component B from T2 to two weeks later (T4), and Component A from T4 to two weeks later (T6). Target n = 7.
  Interventions: Behavioral: Component A; Behavioral: Component B; Behavioral: Component C

INTERVENTIONS:
Behavioral: Component A — All components consist of one online therapist-led session, and 14 daily assignments. In the online session, parents watch an animation clip explaining the technique, and parents perform an exercise guided by the therapist. In the daily assignments, parents reflect on situations in which their child was anxious during the day in which they (could have) applied the technique. If the child was not anxious that day, parents are asked to think about a future or past situation and fill in similar questions.
  Component A focusses on making parents aware of the process of avoidance in children with anxiety, and helps them to identify situations in which they accommodate to the anxiety of their children. Subsequently, a first step that parents can take to reduce accommodation is discussed.
  Other Names: Family Accommodation
  Arms: Condition 12: 0CA; Condition 14: A00; Condition 15: A0B; Condition 16: A0C; Condition 17: AB0; Condition 18: ABC; Condition 19: AC0; Condition 20: ACB; Condition 22: B0A; Condition 24: BA0; Condition 25: BAC; Condition 27: BCA; Condition 29: C0A; Condition 2: 0A0; Condition 31: CA0; Condition 32: CAB; Condition 34: CBA; Condition 3: 00A; Condition 4: 0AB; Condition 5: 0AC; Condition 8: 0BA
Behavioral: Component B — All components consist of one online therapist-led session, and 14 daily assignments. In the online session, parents watch an animation clip explaining the technique, and parents perform an exercise guided by the therapist. In the daily assignments, parents reflect on situations in which their child was anxious during the day in which they (could have) applied the technique. If the child was not anxious that day, parents are asked to think about a future or past situation and fill in similar questions.
  Component B tries to increase parents empathetic reactions to their anxious child. This is done by teaching parents to label the emotion of their children, empathize with the emotion, and communicate confidence in the abilities of their child to face the situation.
  Other Names: Empathetic Reactions
  Arms: Condition 13: 0CB; Condition 15: A0B; Condition 17: AB0; Condition 18: ABC; Condition 20: ACB; Condition 21: B00; Condition 22: B0A; Condition 23: B0C; Condition 24: BA0; Condition 25: BAC; Condition 26: BC0; Condition 27: BCA; Condition 30: C0B; Condition 32: CAB; Condition 33: CB0; Condition 34: CBA; Condition 4: 0AB; Condition 6: 0B0; Condition 7: 00B; Condition 8: 0BA; Condition 9: 0BC
Behavioral: Component C — All components consist of one online therapist-led session, and 14 daily assignments. In the online session, parents watch an animation clip explaining the technique, and parents perform an exercise guided by the therapist. In the daily assignments, parents reflect on situations in which their child was anxious during the day in which they (could have) applied the technique. If the child was not anxious that day, parents are asked to think about a future or past situation and fill in similar questions.
  Component C consists of cognitive restructuring of parental maladaptive cognitions concerning their child's anxiety. Parents are taught to recognize their own cognitions about the anxiety of their child, challenge this thought and come up with an alternative, helpful thought.
  Other Names: Cognitive Restructuring
  Arms: Condition 10: 0C0; Condition 11: 00C; Condition 12: 0CA; Condition 13: 0CB; Condition 16: A0C; Condition 18: ABC; Condition 19: AC0; Condition 20: ACB; Condition 23: B0C; Condition 25: BAC; Condition 26: BC0; Condition 27: BCA; Condition 28: C00; Condition 29: C0A; Condition 30: C0B; Condition 31: CA0; Condition 32: CAB; Condition 33: CB0; Condition 34: CBA; Condition 5: 0AC; Condition 9: 0BC

SUMMARY:
This trial will test the relative effects of three parent-intervention components to reduce emerging anxiety problems in children aged 7-11. The components are: reducing family accommodation (Component A), increasing empathetic reactions to children's anxiety (Component B), and cognitive restructuring to reduce maladaptive parental thoughts about children's anxiety (Component C). The components were selected based on their distinct theoretical backgrounds and their frequent use in existing intervention programs. The investigators will use a full factorial experiment with all possible combinations and orders of components. The study period will be twelve weeks with five points of data-collection: T0 (baseline), T2 (two weeks post baseline, immediately after the first component), T4 (four weeks post baseline, immediately after the second component), T6 (six weeks post baseline, immediately after the third component) and T12 (12 weeks post baseline, follow-up).

Our overarching research questions are:

* How effective are Component A, B, and C in reducing children's anxiety symptoms? The effects of the components will be compared with each other, and with a control condition. This will be investigated both from T0 to T2 (i.e., effects of the individual components) and from T0 to T6 and T0 to T12 (i.e., effects of the components controlled for the presence of other components).
* How effective are the components in reducing children's life impairment? The effects of the components will be compared with each other, and with a control condition.
* Are effects of the components on children's anxiety mediated by changes in the parental risk factors that they target? (i.e., family accommodation for Component A, empathetic reactions for Component B, and parental maladaptive beliefs about child anxiety for Component C)
* Is there a dose-response effect such that children whose parents received more intervention components benefit more in terms of reduced anxiety symptoms in children?
* What parent, child, and intervention characteristics moderate the effects of the components on children's anxiety? In addition to basic sociodemographic information, the investigators will collect data on several putative moderators: the extent to which parents see their child as part of themselves (Inclusion of Child in the Self Scale), children's behavioural inhibition (Behavioural Inhibition Questionnaire), therapist alliance (Session Rating Scale), acceptability of the intervention (TEI-SF), other caregiver's use of the intervention components.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 7;0 - 11;11 years old
* Score of ≥ 4 on the screening questionnaire "Overall Anxiety Severity and Impairment Scale for Youth" (OASIS-Y; Comer et al., 2022) filled in by parents.

Exclusion Criteria:

None

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 266 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Child Anxiety | Baseline (T0)
  Screen for Child Anxiety Related Emotional Disorders-NL Parent-version (71 item version but we omitted OCD and PTSS scale and used the remaining 58 items). Higher scores indicate higher anxiety.
Child Anxiety | Two weeks after baseline (T2)
  Screen for Child Anxiety Related Emotional Disorders-NL Parent-version (71 item version but we omitted OCD and PTSS scale and used the remaining 58 items). Higher scores indicate higher anxiety.
Child Anxiety | Four weeks after baseline (T4)
  Screen for Child Anxiety Related Emotional Disorders-NL Parent-version (71 item version but we omitted OCD and PTSS scale and used the remaining 58 items). Higher scores indicate higher anxiety.
Child Anxiety | Six weeks after baseline (T6)
  Screen for Child Anxiety Related Emotional Disorders-NL Parent-version (71 item version but we omitted OCD and PTSS scale and used the remaining 58 items). Higher scores indicate higher anxiety.
Child Anxiety | Twelve weeks after baseline (T12, follow-up)
  Screen for Child Anxiety Related Emotional Disorders-NL Parent-version (71 item version but we omitted OCD and PTSS scale and used the remaining 58 items). Higher scores indicate higher anxiety.

SECONDARY OUTCOMES:
Child Life impairment | Baseline (T0)
  Child Anxiety Life Interference Scale . Higher scores indicate more life interference.
Child Life impairment | Two weeks after baseline (T2)
  Child Anxiety Life Interference Scale. Higher scores indicate more life interference.
Child Life impairment | Four weeks after baseline (T4)
  Child Anxiety Life Interference Scale. Higher scores indicate more life interference.
Child Life impairment | Six weeks after baseline (T6)
  Child Anxiety Life Interference Scale. Higher scores indicate more life interference.
Child Life impairment | Twelve weeks after baseline (T12, follow-up)
  Child Anxiety Life Interference Scale. Higher scores indicate more life interference.
Family Accommodation | Baseline (T0)
  Family Accommodation Scale - Anxiety. Higher scores indicate more family accommodation.
Family Accommodation | Two weeks after baseline (T2)
  Family Accommodation Scale - Anxiety. Higher scores indicate more family accommodation.
Family Accommodation | Four weeks after baseline (T4)
  Family Accommodation Scale - Anxiety. Higher scores indicate more family accommodation.
Family Accommodation | Six weeks after baseline (T6)
  Family Accommodation Scale - Anxiety. Higher scores indicate more family accommodation.
Family Accommodation | Twelve weeks after baseline (T12, follow-up)
  Family Accommodation Scale - Anxiety. Higher scores indicate more family accommodation.
Parental Empathetic Reactions to Child Anxiety | Baseline (T0)
  Questionnaire loosely based on the Empathy Formative Questionnaire. Higher scores indicate more empathy.
Parental Empathetic Reactions to Child Anxiety | Two weeks after baseline (T2)
  Questionnaire loosely based on the Empathy Formative Questionnaire. Higher scores indicate more empathy.
Parental Empathetic Reactions to Child Anxiety | Four weeks after baseline (T4)
  Questionnaire loosely based on the Empathy Formative Questionnaire. Higher scores indicate more empathy.
Parental Empathetic Reactions to Child Anxiety | Six weeks after baseline (T6)
  Questionnaire loosely based on the Empathy Formative Questionnaire. Higher scores indicate more empathy.
Parental Empathetic Reactions to Child Anxiety | Twelve weeks after baseline (T12, follow-up)
  Questionnaire loosely based on the Empathy Formative Questionnaire. Higher scores indicate more empathy.
Parental Cognitions about Child Anxiety | Baseline (T0)
  Parental Beliefs About Anxiety Questionnaire. Higher scores indicate more maladaptive cognitions.
Parental Cognitions about Child Anxiety | Two weeks after baseline (T2)
  Parental Beliefs About Anxiety Questionnaire. Higher scores indicate more maladaptive cognitions.
Parental Cognitions about Child Anxiety | Four weeks after baseline (T4)
  Parental Beliefs About Anxiety Questionnaire. Higher scores indicate more maladaptive cognitions.
Parental Cognitions about Child Anxiety | Six weeks after baseline (T6)
  Parental Beliefs About Anxiety Questionnaire. Higher scores indicate more maladaptive cognitions.
Parental Cognitions about Child Anxiety | Twelve weeks after baseline (T12, follow-up)
  Parental Beliefs About Anxiety Questionnaire. Higher scores indicate more maladaptive cognitions.

OTHER OUTCOMES:
Child general mental health | Baseline (T0)
  Behavior and Feeling Survey (anxiety scale omitted). Higher scores indicate worse mental health.
Child general mental health | Six weeks after baseline (T6)
  Behavior and Feeling Survey (anxiety scale omitted). Higher scores indicate worse mental health.
Child general mental health | Twelve weeks after baseline (T12, follow-up)
  Behavior and Feeling Survey (anxiety scale omitted). Higher scores indicate worse mental health.
Parental Anxiety | Baseline (T0)
  Anxiety subscale DASS-21. Higher scores indicate more parental anxiety.
Parental Anxiety | Two weeks after baseline (T2)
  Anxiety subscale DASS-21. Higher scores indicate more parental anxiety.
Parental Anxiety | Four weeks after baseline (T4)
  Anxiety subscale DASS-21. Higher scores indicate more parental anxiety.
Parental Anxiety | Six weeks after baseline (T6)
  Anxiety subscale DASS-21. Higher scores indicate more parental anxiety.
Parental Anxiety | Twelve weeks after baseline (T12, follow-up)
  Anxiety subscale DASS-21
Parental self-efficacy | Baseline (T0)
  Self-efficacy subscale Me as a Parent. Higher scores indicate more self-efficacy.
Parental self-efficacy | Two weeks after baseline (T2)
  Self-efficacy subscale Me as a Parent. Higher scores indicate more self-efficacy.
Parental self-efficacy | Four weeks after baseline (T4)
  Self-efficacy subscale Me as a Parent. Higher scores indicate more self-efficacy.
Parental self-efficacy | Six weeks after baseline (T6)
  Self-efficacy subscale Me as a Parent . Higher scores indicate more self-efficacy.
Parental self-efficacy | Twelve weeks after baseline (T12, follow-up)
  Self-efficacy subscale Me as a Parent. Higher scores indicate more self-efficacy.
Parental anxiety change expectancy | Baseline (T0)
  Variation on the Anxiety Change Expectancy Scale. Higher scores indicate more change expectancy.
Parental anxiety change expectancy | Two weeks after baseline (T2)
  Variation on the Anxiety Change Expectancy Scale. Higher scores indicate more change expectancy.
Parental anxiety change expectancy | Four weeks after baseline (T4)
  Variation on the Anxiety Change Expectancy Scale. Higher scores indicate more change expectancy.
Parental anxiety change expectancy | Six weeks after baseline (T6)
  Variation on the Anxiety Change Expectancy Scale. Higher scores indicate more change expectancy.
Parental anxiety change expectancy | Twelve weeks after baseline (T12, follow-up)
  Variation on the Anxiety Change Expectancy Scale. Higher scores indicate more change expectancy.
Parent-child interactions | Baseline (T0)
  Parent-child discussion task with increasing levels of difficulty. The task will be recorded, and coded by independent coders who are blind for the condition of the participants and timepoint of the recording. The observations will be coded for behavior relevant to those behaviors targeted in the intervention components.
Parent-child interactions | Six weeks after baseline (T6)
  Parent-child discussion task with increasing levels of difficulty. The task will be recorded, and coded by independent coders who are blind for the condition of the participants and timepoint of the recording. The observations will be coded for behavior relevant to those behaviors targeted in the intervention components.
Parent-child interactions | Twelve weeks after baseline (T12, follow-up)
  Parent-child discussion task with increasing levels of difficulty. The task will be recorded, and coded by independent coders who are blind for the condition of the participants and timepoint of the recording. The observations will be coded for behavior relevant to those behaviors targeted in the intervention components.
Clinician rated child anxiety | Baseline (T0)
  Secondary clinician rated measure of child anxiety, additionally to the parent report. A verbal interview with the parents will be performed, using the questions of the Overall Anxiety Severity and Impairment Scale for youth (OASIS-Y). The questions will be presented as open-ended questions (i.e., without the original OASIS-Y multiple choice options), and parents are asked to answer freely. This will be recorded, and afterwards the answers will be coded by independent clinicians who will rate the parents' answers using the original OASIS-Y answer categories. Higher scores indicate a worse outcome.
Clinician rated child anxiety | Six weeks after baseline (T6)
  Secondary clinician rated measure of child anxiety, additionally to the parent report. A verbal interview with the parents will be performed, using the questions of the Overall Anxiety Severity and Impairment Scale for youth (OASIS-Y). The questions will be presented as open-ended questions (i.e., without the original OASIS-Y multiple choice options), and parents are asked to answer freely. This will be recorded, and afterwards the answers will be coded by independent clinicians who will rate the parents' answers using the original OASIS-Y answer categories. Higher scores indicate a worse outcome.
Clinician rated child anxiety | Twelve weeks after baseline (T12, follow-up)
  Secondary clinician rated measure of child anxiety, additionally to the parent report. A verbal interview with the parents will be performed, using the questions of the Overall Anxiety Severity and Impairment Scale for youth (OASIS-Y). The questions will be presented as open-ended questions (i.e., without the original OASIS-Y multiple choice options), and parents are asked to answer freely. This will be recorded, and afterwards the answers will be coded by independent clinicians who will rate the parents' answers using the original OASIS-Y answer categories. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Rienks, MSc, Principal Investigator — University of Amsterdam; Patty Leijten, Dr, Study Director — University of Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymized data will be publicly shared after publication of the project results.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After publication of project results
Access Criteria: Via UvA Figshare data can be stored and shared on request. Requests are considered by the study officials. Together they decide whether anonymised data can be shared with a third party.

REFERENCES:
- [Background] Bodden DH, Bogels SM, Muris P. The diagnostic utility of the Screen for Child Anxiety Related Emotional Disorders-71 (SCARED-71). Behav Res Ther. 2009 May;47(5):418-25. doi: 10.1016/j.brat.2009.01.015. Epub 2009 Jan 30. PMID 19230863
- [Background] Lyneham HJ, Sburlati ES, Abbott MJ, Rapee RM, Hudson JL, Tolin DF, Carlson SE. Psychometric properties of the Child Anxiety Life Interference Scale (CALIS). J Anxiety Disord. 2013 Oct;27(7):711-9. doi: 10.1016/j.janxdis.2013.09.008. Epub 2013 Sep 26. PMID 24135256
- [Background] Lebowitz ER, Woolston J, Bar-Haim Y, Calvocoressi L, Dauser C, Warnick E, Scahill L, Chakir AR, Shechner T, Hermes H, Vitulano LA, King RA, Leckman JF. Family accommodation in pediatric anxiety disorders. Depress Anxiety. 2013 Jan;30(1):47-54. doi: 10.1002/da.21998. Epub 2012 Sep 10. PMID 22965863
- [Background] Francis SE, Chorpita BF. Development and Evaluation of the Parental Beliefs about Anxiety Questionnaire. J Psychopathol Behav Assess. 2010;32(1):138-149. doi:10.1007/s10862-009-9133-5
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Lovibond SH, Lovibond PF. Manual for the Depression Anxiety Stress Scales. 2nd ed. Psychology Foundation of Australia; 1995.
- [Background] de Beurs E, Van Dyck R, Marquenie LA, Lange A, Blonk RWB. De DASS: Een vragenlijst voor het meten van depressie, angst en stress. [The DASS: A questionnaire for the measurement of depression, anxiety, and stress.]. Gedragstherapie. 2001;34:35-53.
- [Background] Dozois DJ, Westra HA. Development of the Anxiety Change Expectancy Scale (ACES) and validation in college, community, and clinical samples. Behav Res Ther. 2005 Dec;43(12):1655-72. doi: 10.1016/j.brat.2004.12.001. PMID 15922290
- [Background] van der Sterren-Kusters WJC, van der Heijden PT, Egger JIM. Psychometric Properties of the Dutch Anxiety Change Expectancy Scale (ACES-NL). Int J Psychol Psychol Ther. 2017;17:189-198.
- [Background] Aron A, Aron EN, Smollan D. Inclusion of Other in the Self Scale and the structure of interpersonal closeness. J Pers Soc Psychol. 1992;63:596-612. doi:10.1037/0022-3514.63.4.596
- [Background] Brummelman E, Thomaes S, Slagt M, Overbeek G, de Castro BO, Bushman BJ. My Child Redeems My Broken Dreams: On Parents Transferring Their Unfulfilled Ambitions onto Their Child. PLoS One. 2013 Jun 19;8(6):e65360. doi: 10.1371/journal.pone.0065360. Print 2013. PMID 23840325
- [Background] Bishop G, Spence SH, McDonald C. Can parents and teachers provide a reliable and valid report of behavioral inhibition? Child Dev. 2003 Nov-Dec;74(6):1899-917. doi: 10.1046/j.1467-8624.2003.00645.x. PMID 14669903
- [Background] Duncan BL, Miller SD, Sparks JA, et al. The Session Rating Scale: Preliminary Psychometric Properties of a "Working" Alliance Measure. J Brief Ther. 2003;3(1):3-12.
- [Background] Kazdin AE. Acceptability of child treatment techniques: The influence of treatment efficacy and adverse side effects. Behav Ther. 1981;12(4):493-506. doi:10.1016/S0005-7894(81)80087-1
- [Background] Kelley ML, Heffer RW, Gresham FM, Elliott SN. Development of a modified treatment evaluation inventory. J Psychopathol Behav Assess. 1989;11(3):235-247. doi:10.1007/BF00960495
- [Background] Hamilton VE, Matthews JM, Crawford SB. Me as a Parent Questionnaire [Database record]. APA PsycTests. 2015. doi:10.1037/t45911-000
- [Background] Gaumer Erickson AS, Soukup JH, Noonan PM, McGurn L. Empathy Formative Questionnaire. College & Career Competency Framework. 2015. https://www.cccframework.org/
- [Background] Comer JS, Conroy K, Cornacchio D, Furr JM, Norman SB, Stein MB. Psychometric evaluation of a caregiver-report adaptation of the Overall Anxiety Severity and Impairment Scale (OASIS) for use with youth populations. J Affect Disord. 2022 Mar 1;300:341-348. doi: 10.1016/j.jad.2021.12.113. Epub 2021 Dec 31. PMID 34979182